CLINICAL TRIAL: NCT04477369
Title: An Exploratory Clinical Trial to Compare and Evaluate Safety and Pharmacokinetic Characteristics After Administration of the DWJ1439, DWJ1464, DWC202003 or DWC202004 in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetics of DWJ1439, DWJ1464, DWC202003 or DWC202004 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1464101
Record Dates: First submitted 2020-06-22; First posted 2020-07-20 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence A (Other): 7 subjects assigned to Sequence A will receive a single dose of 300mg DWJ1439 in period 1, 300mg DWC202003 in period 2 and 300mg DWJ1464 in period 3.
  Interventions: Drug: DWJ1439; Drug: DWJ1464; Drug: DWC202003
- Sequence B (Other): 7 subjects assigned to Sequence B will receive a single dose of 300mg DWJ1464 in period 1, 300mg DWC202004 in period 2 and 300mg DWC202003 in period 3.
  Interventions: Drug: DWJ1464; Drug: DWC202003; Drug: DWC202004
- Sequence C (Other): 7 subjects assigned to Sequence C will receive a single dose of 300mg DWC202003 in period 1, 300mg DWJ1439 in period 2 and 300mg DWC202004 in period 3.
  Interventions: Drug: DWJ1439; Drug: DWC202003; Drug: DWC202004
- Sequence D (Other): 7 subjects assigned to Sequence D will receive a single dose of 300mg DWC202004 in period 1, 300mg DWJ1464 in period 2 and 300mg DWJ1439 in period 3.
  Interventions: Drug: DWJ1439; Drug: DWJ1464; Drug: DWC202004

INTERVENTIONS:
Drug: DWJ1439 — 300mg single dose
  Arms: Sequence A; Sequence C; Sequence D
Drug: DWJ1464 — 300mg single dose
  Arms: Sequence A; Sequence B; Sequence D
Drug: DWC202003 — 300mg single dose
  Arms: Sequence A; Sequence B; Sequence C
Drug: DWC202004 — 300mg single dose
  Arms: Sequence B; Sequence C; Sequence D

SUMMARY:
The purpose of this study is to explore the differences in pharmacokinetics and safety characteristics between Test Drugs(DWJ1439, DWJ1464) and that of Reference Drugs(DWC202003, DWC202004) in healthy adults.

DETAILED DESCRIPTION:
The purpose of this study is to explore the differences in pharmacokinetics and safety characteristics between Test Drugs(DWJ1439, DWJ1464) and that of Reference Drugs(DWC202003, DWC202004) in healthy adults with fasting state: Randomized, open-label, oral, single-dose, four-treatment, three-period, non-replicated crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 years old to under 55.
* BMI 18.0≥ and ≤30 kg/m² with body mass ≥50 kg
* Those who have no congenital or chronic disease requiring treatment and have no pathological symptoms or findings as a result of medical examination.
* Those who have no clinically significant abnormalities in general physical examination, laboratory assessments and 12-lead electrocardiogram (ECG).
* Those who understand the requirements of the study and sign a written informed consent, and also accept all the restrictions imposed during the course of the study.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Participation in a clinical drug study or bioequivalence study 6 months prior to the present study.
* Refusal to abstain from smoking or consumption of tobacco products 72 hours before drug administration and during each study period.
* Refusal to abstain from alcohol, caffeine, or other xanthines, or grapefruit containing food or drinks for 72 hours before drug administration and during each study period.
* Refusal to abstain from strenuous activities for 72 hours before drug administration and post-study visit, before and during each study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-08-06 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: AUC0-t | 0 - 72 hours after dosing
  Area under the plasma concentration-time curve from time 0 to time t
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: Cmax | 0 - 72 hours after dosing
  Maximum plasma drug concentration
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: AUC0-t | 0 - 72 hours after dosing
  Area under the plasma concentration-time curve from time 0 to time t
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: Cmax | 0 - 72 hours after dosing
  Maximum plasma drug concentration

SECONDARY OUTCOMES:
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: AUCinf | 0 - 72 hours after dosing
  Area under the plasma concentration-time curve from drug administration to drug elimination
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: Tmax | 0 - 72 hours after dosing
  Time to reach maximum plasma concentration following drug administration
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: t1/2 | 0 - 72 hours after dosing
  Elimination half-life
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: , Cl/F | 0 - 72 hours after dosing
  Apparent total clearance of drug from plasma after oral administration
PK parameters of baseline corrected/uncorrected ursodeoxycholic acid: Vd/F | 0 - 72 hours after dosing
  Apparent volume of distribution after oral administration
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: AUCinf | 0 - 72 hours after dosing
  Area under the plasma concentration-time curve from drug administration to drug elimination
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: Tmax | 0 - 72 hours after dosing
  Time to reach maximum plasma concentration following drug administration
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: t1/2 | 0 - 72 hours after dosing
  Elimination half-life
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: Cl/F | 0 - 72 hours after dosing
  Apparent total clearance of drug from plasma after oral administration
PK parameters of baseline corrected/uncorrected total ursodeoxycholic acid: Vd/F | 0 - 72 hours after dosing
  Apparent volume of distribution after oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Medical Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No